CLINICAL TRIAL: NCT03366831
Title: Thirty Million Words Initiative Newborn Implementation Trial
Brief Title: Newborn Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17-0329
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Language Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15 minute version without questions (Active Comparator): 15 minute version of the TMW-Newborn intervention video without questions interspersed
  Interventions: Behavioral: Thirty Million Words Initiative Newborn Intervention
- 15 minute version with questions (Active Comparator): 15 minute version of the TMW-Newborn intervention video with questions interspersed
  Interventions: Behavioral: Thirty Million Words Initiative Newborn Intervention
- 7 minute version without questions (Active Comparator): 7 minute version of the TMW-Newborn intervention video without questions interspersed
  Interventions: Behavioral: Thirty Million Words Initiative Newborn Intervention
- 7 minute version with questions (Active Comparator): 7 minute version of the TMW-Newborn intervention video with questions interspersed.
  Interventions: Behavioral: Thirty Million Words Initiative Newborn Intervention

INTERVENTIONS:
Behavioral: Thirty Million Words Initiative Newborn Intervention — The Thirty Million Words Initiative Newborn Intervention (TMW-Newborn) is a public health effort aimed at increasing awareness about the importance of a child's early language environment in his or her first years of life. This one-time educational intervention will be impacting maternal awareness and knowledge about the importance of children's early language environment, between ages 0 and 3.

SUMMARY:
The purpose of the proposed research is to perform testing of the Thirty Million Words Newborn Initiative (TMW-NI) with the primary goal of evaluating various implementation methods.

The investigators hypothesize that the TMW-Newborn intervention will:

1. Significantly impact parent knowledge regarding the importance of universal newborn hearing screen (UNHS) follow-up
2. Significantly impact parent knowledge of child development

   Additionally,the investigators hypothesize that:
3. The 7-minute version of the video with questions interspersed will most significantly improve parent knowledge of child development
4. There will be no significant differences in effectiveness of the Spanish and English versions of the TMW-Newborn intervention

The hypotheses rely on the existing research data supporting the idea that parental understanding and beliefs will alter parental behavior, and consequently, that increased parental linguistic input will impact child cognitive development.

DETAILED DESCRIPTION:
The investigators propose to perform a randomized implementation trial to evaluate the efficacy of various implementation methods of the TMW-Newborn educational intervention. The study will be conducted in temporal proximity to the administration of the universal newborn hearing screen.

After routine delivery, postpartum mothers are admitted to the mother-baby unit for 48-72 hours. A hearing screening technician of the Sacred Heart Hospital will deliver the tablet that houses the intervention to every mother whose child is receiving the hearing screening. The technician will give each mother a tablet set up to the HIPAA Compliant TMW-Newborn Web Platform that houses the randomization tool, the welcome video, the tablet based consent passage, the surveys, and the educational intervention videos. First, the participant will watch the welcome video and complete the tablet based consent. Then, the participant will be randomized into one of four conditions: 15 minute version of the TMW-Newborn intervention video without questions interspersed, the 15 minute version of the TMW-Newborn intervention video with questions interspersed, the 7 minute version of the TMW-Newborn intervention video without questions interspersed, or the 7 minute version of the TMW-Newborn intervention video with questions interspersed.

After randomization, the participant will be brought to the screen with the SPEAK III to complete. Then, they will answer a few non-identifying demographics questions. These surveys takes approximately 10 minutes to complete will be followed by either a 15-minute or 7-minute video.

After watching their assigned video, all participants will repeat the SPEAK questionnaire for a second time. Then, the hearing screener will pick up the tablet from the participant. No identifying information is being collected within the TMW-Newborn web platform, and the hearing screening technicians will not be able to see or access any of the participants' responses.

After all surveys are complete, the hearing screening technician will pick up the tablet from the participant and answer any remaining questions.

This study protocol will only be used at Sacred Heart Hospital, Baptist Hospital, and University of Chicago Hospital.

ELIGIBILITY:
Inclusion Criteria:

New mothers at Sacred Heart Hospital, University of Chicago Medical Center, and Baptist Hospital-Pensacola.

Exclusion Criteria:

Individuals that do not have a live birth at Sacred Heart Hospital, University of Chicago Medical Center, or Baptist Hospital-Pensacola or do not receive the UNHS at one of these locations will not be eligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — new mothers
Enrollment: 2701 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
SPEAK Survey (Baby Subscales) | 48-72 after routine delivery
  measures an individuals expectations and knowledge about child development

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sacred Heart Hospital, Pensacola, Florida
  - Baptist Hospital, Pensacola, Florida
  - TMW Center for Early Learning + Public Health at the University of Chicago Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Suskind DL, Leung CYY, Webber RJ, Hundertmark AC, Leffel KR, Fuenmayor Rivas IE, Grobman WA. Educating Parents About Infant Language Development: A Randomized Controlled Trial. Clin Pediatr (Phila). 2018 Jul;57(8):945-953. doi: 10.1177/0009922817737079. Epub 2017 Oct 26. PMID 29073768
- See also: Click here for more information about the Thirty Million Words — https://tmwcenter.uchicago.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03366831/Prot_SAP_000.pdf